CLINICAL TRIAL: NCT04200651
Title: Prospective Study on DEXTENZA® Safety And Efficacy Following Concomitant MIGS and Cataract Surgery
Acronym: SUSTAIN
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID-19 challenges to recruitment
Sponsor: The New York Eye Surgery Center (Other)
Collaborators: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Principal Investigator, Nathan M. Radcliffe, MD, Dr. Nathan M. Radcliffe, Attending Ophthalmologist, The New York Eye Surgery Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 146602
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Results first posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Glaucoma; Cataract
Keywords: MIGS, Minimally invasive glaucoma surgery
MeSH Terms: conditions — Glaucoma; Cataract | interventions — Calcium Dobesilate; prednisolone acetate; Methylprednisolone

STUDY DESIGN:
Intervention Model Description: This prospective study enrolled 29 eyes from 25 total patients. The protocol permitted some binocular enrollment from patients who met eligibility criteria in both eyes.
  All eligible eyes received concomitant cataract and MIGS surgery. Each eye was randomized to receive either DEXTENZA® insertion at the end of the surgery or to a standard of care prednisolone acetate 1% eye drop regimen via block randomization. All eyes received the standard of care topical ofloxacin antibiotic regimen. The experimental group consisted of the eyes receiving DEXTENZA® insertion. The control group consisted of the eyes placed on the prednisolone eye drop regimen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DEXTENZA® arm (Experimental): This arm will receive the DEXTENZA® insert after cataract surgery and MIGS.
  Interventions: Drug: Dexamethasone Ophthalmic Insert
- Prednisolone acetate 1% arm (Active Comparator): This arm will receive the prescription for daily prednisolone acetate 1% eye drops after cataract surgery and MIGS.
  Interventions: Drug: Prednisolone Acetate 1% Oph Susp

INTERVENTIONS:
Drug: Dexamethasone Ophthalmic Insert — DEXTENZA® is a 3mm long gel-like cylinder that is inserted in the punctum, a natural opening in the lower eyelid. DEXTENZA® is activated by the eye's moisture. DEXTENZA® delivers 0.4 mg dexamethasone, a liquid corticosteroid, onto the surface of the eye automatically for up to 30 days after eye surgery. Dexamethasone is used to reduce inflammation and eye pain. This arm will also receive the standard of care topical ofloxacin eye drop antibiotic regimen.
  Other Names: DEXTENZA®
  Arms: DEXTENZA® arm
Drug: Prednisolone Acetate 1% Oph Susp — Prednisolone acetate 1% eye drops are used 2-4 times daily for 30 days as the current standard of care for treating inflammation and eye pain after cataract surgery. Prednisolone, like dexamethasone, is a steroid. This arm will also receive the standard of care topical ofloxacin eye drop antibiotic regimen.
  Other Names: PRED FORTE®, OMNIPRED®
  Arms: Prednisolone acetate 1% arm

SUMMARY:
In this study, the investigators are comparing dexamethasone ophthalmic insert (DEXTENZA®) to the current standard of care, prednisolone acetate 1% eye drops, in a glaucoma population receiving both cataract and minimally-invasive glaucoma surgery (MIGS). DEXTENZA® and prednisolone acetate 1% drops are both steroids used to control inflammation after eye surgery. DEXTENZA®'s method of delivery differs by offering a sustained release of steroid that does not necessitate postoperative anti-inflammatory eye drops. The investigators hypothesize that DEXTENZA® will be as safe as prednisolone acetate 1% drops and as effective at controlling postoperative inflammation following concomitant cataract-MIGS in a glaucoma population. The investigators also hypothesize that DEXTENZA® will be preferred by patients over prednisolone acetate 1% drops.

DETAILED DESCRIPTION:
Glaucoma and cataract surgery patients face an outsize postoperative burden. In addition to taking frequent anti-inflammatory eye drops, they often continue their glaucoma medications. This can cause patient confusion and nonadherence, potentially leading to poor healing, slower recovery period, and/or cystoid macular edema. DEXTENZA®, as a sustained release anti-inflammatory insert, could help preclude adherence difficulties and increase comfort by reducing eye drop load. However, glaucoma surgeons may hesitate to adopt DEXTENZA® due to concerns regarding safety with respect to elevated intraocular pressure. This prospective study will address those concerns directly, providing timely and high-quality clinical evidence comparing DEXTENZA® to standard-of-care steroid eye drops. For physicians and patients, the results of this study will prove immediately useful for therapeutic decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Cataract surgery candidate and glaucoma present in at least one eye.
* Minimally-invasive glaucoma surgery candidate in that same eye. Defined by having ocular hypertension requiring a medication, OR as by having mild, moderate, or severe glaucoma that is sufficiently stable and appropriate for operation.

Exclusion Criteria:

* Maintains regular use (daily or more) of systemic or ocular steroids at time of enrollment
* Maintains regular use (daily or more) of systemic or ocular nonsteroidal anti-inflammatory drugs at time of enrollment
* Anterior chamber cells present at time of enrollment
* Recent febrile illness that precludes or delays participation for 3 months
* Pregnancy or lactation
* Known allergy to dexamethasone
* Known allergy to prednisolone
* Treatment with another investigational drug within the last 20 years
* Current recreational drug use
* Preexisting ocular pathology likely to confound the visual acuity or comfort endpoints including but not limited to: severe corneal scarring, ocular surface disease, diabetic retinopathy, or macular edema
* Corneal or retinal procedures (laser or incisional) during the study period and 6 months prior

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan M Radcliffe, MD, Principal Investigator — New York Eye Surgery Center; New York Eye and Ear Infirmary of Mount Sinai
Locations (1):
- The New York Eye Surgery Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Johnson ME, Murphy PJ. Measurement of ocular surface irritation on a linear interval scale with the ocular comfort index. Invest Ophthalmol Vis Sci. 2007 Oct;48(10):4451-8. doi: 10.1167/iovs.06-1253. PMID 17898265
- [Background] Juthani VV, Clearfield E, Chuck RS. Non-steroidal anti-inflammatory drugs versus corticosteroids for controlling inflammation after uncomplicated cataract surgery. Cochrane Database Syst Rev. 2017 Jul 3;7(7):CD010516. doi: 10.1002/14651858.CD010516.pub2. PMID 28670710
- [Background] Kindle T, Ferguson T, Ibach M, Greenwood M, Schweitzer J, Swan R, Sudhagoni RG, Berdahl JP. Safety and efficacy of intravitreal injection of steroid and antibiotics in the setting of cataract surgery and trabecular microbypass stent. J Cataract Refract Surg. 2018 Jan;44(1):56-62. doi: 10.1016/j.jcrs.2017.10.040. PMID 29502618
- [Background] Newman-Casey PA, Robin AL, Blachley T, Farris K, Heisler M, Resnicow K, Lee PP. The Most Common Barriers to Glaucoma Medication Adherence: A Cross-Sectional Survey. Ophthalmology. 2015 Jul;122(7):1308-16. doi: 10.1016/j.ophtha.2015.03.026. Epub 2015 Apr 24. PMID 25912144
- [Background] Fisher BL, Potvin R. Transzonular vitreous injection vs a single drop compounded topical pharmaceutical regimen after cataract surgery. Clin Ophthalmol. 2016 Jul 18;10:1297-303. doi: 10.2147/OPTH.S112080. eCollection 2016. PMID 27486301

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total, 25 subjects contributing 29 eyes were consented for the study. Of those 29 eyes consented, 5 eyes from 5 subjects met exclusion criteria, thus leaving 24 eyes from 20 subjects who started the study as described below.
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | DEXTENZA® Arm | Prednisolone Acetate 1% Arm
Started | 14; 14 Eyes | 10; 10 Eyes
Completed | 11; 11 Eyes | 5; 5 Eyes
Not Completed | 3; 3 Eyes | 5; 5 Eyes
Not completed — Moved to another country during follow-up | 2 | 2
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Population: 24 eyes from 20 subjects were consented and met criteria for the study (see Participant Flow Overview). However, prior to full baseline assessment and prior to surgery, 6 eyes from 4 subjects dropped out, leaving 18 eyes from 16 subjects. Additionally, given that a mixed-eye sample can impact statistical assumptions of independence, baseline data comparisons were separated between single eyes and fellow-eyes.
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | DEXTENZA® Arm | Prednisolone Acetate 1% Arm | Total
Number analyzed (Participants) | 12 | 6 | 16
Number analyzed (Eyes) | 12 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Rows have been split into single eyes (eyes from individual participants) and fellow-eyes (eyes from the same participants).
  years
    Single eyes: number analyzed (Participants) | 10 | 4 | 14
    Single eyes: number analyzed (Eyes) | 10 | 4 | 14
    Single eyes | 70.6 (11.65) | 73 (6.32) | 71.3 (10.22)
    Fellow eyes: number analyzed (Participants) | 2 | 2 | 2
    Fellow eyes: number analyzed (Eyes) | 2 | 2 | 4
    Fellow eyes | 67 (9.90) | 67 (9.90) | 67 (8.08)
Sex: Female, Male [Count of Units; unit: Eyes] — Population: Rows have been split into single eyes (eyes from individual participants) and fellow-eyes (eyes from the same participants).
  Eyes
    Single eyes: number analyzed (Participants) | 10 | 4 | 14
    Single eyes: number analyzed (Eyes) | 10 | 4 | 14
    Single eyes: Female | 5 | 3 | 8
    Single eyes: Male | 5 | 1 | 6
    Fellow eyes: number analyzed (Participants) | 2 | 2 | 2
    Fellow eyes: number analyzed (Eyes) | 2 | 2 | 4
    Fellow eyes: Female | 2 | 2 | 4
    Fellow eyes: Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Units; unit: Eyes] — Population: Rows have been split into single eyes (eyes from individual participants) and fellow-eyes (eyes from the same participants).
  Eyes
    Single eyes: number analyzed (Participants) | 10 | 4 | 14
    Single eyes: number analyzed (Eyes) | 10 | 4 | 14
    Single eyes: Asian | 1 | 0 | 1
    Single eyes: Black | 2 | 1 | 3
    Single eyes: White | 1 | 1 | 2
    Single eyes: Hispanic/Latino | 6 | 2 | 8
    Fellow eyes: number analyzed (Participants) | 2 | 2 | 2
    Fellow eyes: number analyzed (Eyes) | 2 | 2 | 4
    Fellow eyes: Asian | 0 | 0 | 0
    Fellow eyes: Black | 2 | 2 | 4
    Fellow eyes: White | 0 | 0 | 0
    Fellow eyes: Hispanic/Latino | 0 | 0 | 0
Region of Enrollment [Number; unit: Eyes]
  United States | 12 | 6 | 18
Prior glaucoma laser treatment [Count of Units; unit: Eyes] — Population: Rows have been split into single eyes (eyes from individual participants) and fellow-eyes (eyes from the same participants).
  Eyes
    Single eyes: number analyzed (Participants) | 10 | 4 | 14
    Single eyes: number analyzed (Eyes) | 10 | 4 | 14
    Single eyes | 3 | 0 | 3
    Fellow eyes: number analyzed (Participants) | 2 | 2 | 2
    Fellow eyes: number analyzed (Eyes) | 2 | 2 | 4
    Fellow eyes | 2 | 2 | 4
Minimally invasive glaucoma surgery (MIGS) type [Count of Units; unit: Eyes] — Population: Rows have been split into single eyes (eyes from individual participants) and fellow-eyes (eyes from the same participants).
  Eyes
    Single eyes: number analyzed (Participants) | 10 | 4 | 14
    Single eyes: number analyzed (Eyes) | 10 | 4 | 14
    Single eyes: Hydrus | 2 | 2 | 4
    Single eyes: iStent | 1 | 0 | 1
    Single eyes: Canaloplasty | 7 | 2 | 9
    Fellow eyes: number analyzed (Participants) | 2 | 2 | 2
    Fellow eyes: number analyzed (Eyes) | 2 | 2 | 4
    Fellow eyes: Hydrus | 1 | 1 | 2
    Fellow eyes: iStent | 0 | 0 | 0
    Fellow eyes: Canaloplasty | 1 | 1 | 2
Glaucoma severity [Count of Units; unit: Eyes] — Population: Rows have been split into single eyes (eyes from individual participants) and fellow-eyes (eyes from the same participants).
  Eyes
    Single eyes: number analyzed (Participants) | 10 | 4 | 14
    Single eyes: number analyzed (Eyes) | 10 | 4 | 14
    Single eyes: Mild glaucoma | 0 | 0 | 0
    Single eyes: Moderate glaucoma | 10 | 4 | 14
    Fellow eyes: number analyzed (Participants) | 2 | 2 | 2
    Fellow eyes: number analyzed (Eyes) | 2 | 2 | 4
    Fellow eyes: Mild glaucoma | 0 | 1 | 1
    Fellow eyes: Moderate glaucoma | 2 | 1 | 3
Intraocular pressure (IOP) [Mean (Standard Deviation); unit: mmHg] — Population: Rows have been split into single eyes (eyes from individual participants) and fellow-eyes (eyes from the same participants).
  mmHg
    Single eyes: number analyzed (Participants) | 10 | 4 | 14
    Single eyes: number analyzed (Eyes) | 10 | 4 | 14
    Single eyes | 17.75 (1.96) | 18.75 (4.86) | 18.04 (2.89)
    Fellow eyes: number analyzed (Participants) | 2 | 2 | 2
    Fellow eyes: number analyzed (Eyes) | 2 | 2 | 4
    Fellow eyes | 16 (5.66) | 16 (5.66) | 16 (4.62)
LogMAR visual acuity [Mean (Standard Deviation); unit: logMAR] — Population: Rows have been split into single eyes (eyes from individual participants) and fellow-eyes (eyes from the same participants).
  logMAR
    Single eyes: number analyzed (Participants) | 10 | 4 | 14
    Single eyes: number analyzed (Eyes) | 10 | 4 | 14
    Single eyes | 0.83 (0.68) | 0.58 (0.30) | 0.76 (0.60)
    Fellow eyes: number analyzed (Participants) | 2 | 2 | 2
    Fellow eyes: number analyzed (Eyes) | 2 | 2 | 4
    Fellow eyes | 0.52 (0.03) | 0.47 (0.10) | 0.50 (0.07)
Central corneal thickness [Mean (Standard Deviation); unit: microns] — Population: Rows have been split into single eyes (eyes from individual participants) and fellow-eyes (eyes from the same participants).
  microns
    Single eyes: number analyzed (Participants) | 10 | 4 | 14
    Single eyes: number analyzed (Eyes) | 10 | 4 | 14
    Single eyes | 521.70 (39.88) | 534.80 (23.39) | 525.44 (35.57)
    Fellow eyes: number analyzed (Participants) | 2 | 2 | 2
    Fellow eyes: number analyzed (Eyes) | 2 | 2 | 4
    Fellow eyes | 492 (5.66) | 475 (4.24) | 483.5 (10.63)
Retinal nerve fiber layer (RNFL) thickness [Mean (Standard Deviation); unit: microns] — Population: Rows have been split into single eyes (eyes from individual participants) and fellow-eyes (eyes from the same participants).
  microns
    Single eyes: number analyzed (Participants) | 10 | 4 | 14
    Single eyes: number analyzed (Eyes) | 10 | 4 | 14
    Single eyes | 72.9 (11.73) | 75.75 (17.29) | 73.71 (12.89)
    Fellow eyes: number analyzed (Participants) | 2 | 2 | 2
    Fellow eyes: number analyzed (Eyes) | 2 | 2 | 4
    Fellow eyes | 53.5 (7.78) | 75 (2.83) | 64.25 (13.3)
Cup-to-disc ratio [Mean (Standard Deviation); unit: ratio] — Anatomic ratio of cup size to disc size as determined on exam, with larger ratios generally correlating with glaucoma severity Population: Rows have been split into single eyes (eyes from individual participants) and fellow-eyes (eyes from the same participants).
  ratio
    Single eyes: number analyzed (Participants) | 10 | 4 | 14
    Single eyes: number analyzed (Eyes) | 10 | 4 | 14
    Single eyes | 0.65 (0.09) | 0.67 (0.07) | 0.66 (0.08)
    Fellow eyes: number analyzed (Participants) | 2 | 2 | 2
    Fellow eyes: number analyzed (Eyes) | 2 | 2 | 4
    Fellow eyes | 0.63 (0.21) | 0.49 (0.20) | 0.56 (0.19)
Glaucoma medications [Mean (Standard Deviation); unit: medications] — Population: Rows have been split into single eyes (eyes from individual participants) and fellow-eyes (eyes from the same participants).
  medications
    Single eyes: number analyzed (Participants) | 10 | 4 | 14
    Single eyes: number analyzed (Eyes) | 10 | 4 | 14
    Single eyes | 1.8 (0.92) | 1.5 (0.58) | 1.7 (0.83)
    Fellow eyes: number analyzed (Participants) | 2 | 2 | 2
    Fellow eyes: number analyzed (Eyes) | 2 | 2 | 4
    Fellow eyes | 1 (0) | 1 (0) | 1 (0)
Visual field mean deviation (VFMD) [Mean (Standard Deviation); unit: dB] — VFMD is an aggregate measure of one's visual field deficits obtained on the Humphrey Visual Field 24-2 algorithm. Generally, more negative values correlate with worse deficits Population: Rows have been split into single eyes (eyes from individual participants) and fellow-eyes (eyes from the same participants).
  dB
    Single eyes: number analyzed (Participants) | 10 | 4 | 14
    Single eyes: number analyzed (Eyes) | 10 | 4 | 14
    Single eyes | -8.45 (4.31) | -4.20 (4.89) | -7.24 (4.73)
    Fellow eyes: number analyzed (Participants) | 2 | 2 | 2
    Fellow eyes: number analyzed (Eyes) | 2 | 2 | 4
    Fellow eyes | -4.74 (NA) — n=1 for VFMD in this group | -2.55 (NA) — n=1 for VFMD in this group | -3.65 (1.10)

OUTCOME MEASURES:

1. Primary Outcome: Change in Intraocular Pressure (IOP) at 1 and 3 Months
Description: Using quantitative IOP readings to compare ocular safety between arms. Since the outcome examined was a "change," baseline, month 1 postop, and month 3 postop data were used in the calculations.
  1 month change calculation: Month 1 postop value - Baseline value 3 month change calculation: Month 3 postop value - Baseline value
Time Frame: 1 month postop, 3 months postop
Population: Change in IOP from baseline at months 1 and 3 were compared between groups.
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: Eyes
Arm/Group | DEXTENZA® Arm | Prednisolone Acetate 1% Arm
Number analyzed (Participants) | 11 | 5
Number analyzed (Eyes) | 11 | 5
mmHg
  Change in IOP by Month 1: number analyzed (Participants) | 9 | 5
  Change in IOP by Month 1: number analyzed (Eyes) | 9 | 5
  Change in IOP by Month 1 | -2.89 (2.37) | -6.60 (3.29)
  Change in IOP by Month 3 | -2.05 (3.30) | -4.6 (3.29)

2. Primary Outcome: Change in Best-corrected Visual Acuity (BCVA) at 1 and 3 Months
Description: Using quantitative BCVA measurements, as determined by ETDRS chart at 4 meters, to compare ocular safety and effectiveness between arms. Since the outcome examined was a "change," baseline, month 1 postop, and month 3 postop data were used in the calculations.
  1 month change calculation: Month 1 postop value - Baseline value 3 month change calculation: Month 3 postop value - Baseline value
Time Frame: 1 month postop, 3 months postop
Population: LogMAR visual acuity changes from baseline to months 1 and 3 were compared between groups. Please note that for logMAR, lower values on the scale correspond with better visual acuity.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | DEXTENZA® Arm | Prednisolone Acetate 1% Arm
Number analyzed (Participants) | 11 | 5
Number analyzed (Eyes) | 11 | 5
logMAR
  LogMAR change by Month 1: number analyzed (Participants) | 9 | 5
  LogMAR change by Month 1: number analyzed (Eyes) | 9 | 5
  LogMAR change by Month 1 | -0.60 (0.63) | -0.16 (0.21)
  LogMAR change by Month 3 | -0.53 (0.66) | -0.20 (0.31)

3. Primary Outcome: Difference in Eyes With Adverse Events Between Groups
Description: Using the average number of eyes with adverse events that occur in each arm to compare safety between arms through 3 months of postoperative follow-up
Time Frame: Up to 3 months postop
Measure: Number; unit: Number of eyes with adverse events
Units Other Than Participants: Eyes
Arm/Group | DEXTENZA® Arm | Prednisolone Acetate 1% Arm
Number analyzed (Participants) | 12 | 6
Number analyzed (Eyes) | 12 | 6
Number of eyes with adverse events | 3 | 0

4. Primary Outcome: Difference in Number of Glaucoma Medications at 3 Months
Description: Using the average number of glaucoma medications added or subtracted to each arm to compare safety between arms. These calculations were performed by subtracting the baseline glaucoma medications from the glaucoma medications at month 3.
Time Frame: 3 months postop
Population: Change in number of glaucoma medications between groups from baseline to month 3 were compared.
Measure: Mean (Standard Deviation); unit: number of medications
Units Other Than Participants: Eyes
Arm/Group | DEXTENZA® Arm | Prednisolone Acetate 1% Arm
Number analyzed (Participants) | 11 | 5
Number analyzed (Eyes) | 11 | 5
number of medications | -0.45 (0.69) | -0.60 (0.89)

5. Secondary Outcome: Percentage of Eyes Requiring Supplemental Prednisolone Acetate 1% Eye Drops
Description: Recording the percentage of eyes in the DEXTENZA® arm that require anti-inflammatory rescue with supplemental ocular steroid. This will provide insight into anti-inflammatory effectiveness of DEXTENZA®
Time Frame: Up to 3 months postop
Population: Of the 14 consented eyes in the DEXTENZA arm noted in the "started" row of the participant flow data table, 2 eyes met exclusion criteria, thus leaving 12 eligible eyes for further analysis.
Measure: Number; unit: Percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | DEXTENZA® Arm
Number analyzed (Participants) | 12
Number analyzed (Eyes) | 12
Percentage of eyes | 25

6. Secondary Outcome: Number of Eyes With Presenting With Cystoid Macular Edema (CME) as Seen on Optical Coherence Tomography (OCT)
Description: Using the number of CME cases in each arm, as visualized by OCT, to compare safety and effectiveness between arms
Time Frame: 3 months postop
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | DEXTENZA® Arm | Prednisolone Acetate 1% Arm
Number analyzed (Participants) | 11 | 5
Number analyzed (Eyes) | 11 | 5
Eyes | 0 | 0

7. Secondary Outcome: Difference in Ocular Comfort Index (OCI) Score at 1 Month
Description: Using the Ocular Comfort Index survey to compare patients' self-reported ocular comfort between arms, providing insight into drug effectiveness. The minimum score is 0 and the maximum score is 100, with 100 indicating the most ocular irritation and discomfort and 0 indicating the least ocular irritation and discomfort
Time Frame: 1 month postop
Population: Scores were compared between groups at month 1. Higher scores correspond to greater ocular discomfort. Of the 18 eyes that received baseline analysis and surgery, only 10 completed the month 1 OCI survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | DEXTENZA® Arm | Prednisolone Acetate 1% Arm
Number analyzed (Participants) | 8 | 2
Number analyzed (Eyes) | 8 | 2
score on a scale | 25.96 (12.50) | 10.71 (15.15)

8. Secondary Outcome: Difference in Ocular Comfort Index (OCI) Score at 3 Months
Description: as for outcome 7
Time Frame: 3 months postop
Population: Scores were compared between groups at month 3. Higher scores correspond to greater ocular discomfort.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | DEXTENZA® Arm | Prednisolone Acetate 1% Arm
Number analyzed (Participants) | 11 | 5
Number analyzed (Eyes) | 11 | 5
score on a scale | 21.20 (14.67) | 16.32 (16.49)

9. Secondary Outcome: Difference in Number of Eyes With Absence of Anterior Chamber (AC) Cells at 1 Month
Description: Comparing the number of eyes with complete AC clearance of inflammatory cells, as determined by slit lamp exam, between arms to evaluate drug effectiveness
Time Frame: 1 month postop
Population: Counts indicate the number of eyes with no AC cell or flare present at 1 month follow-up.
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | DEXTENZA® Arm | Prednisolone Acetate 1% Arm
Number analyzed (Participants) | 9 | 5
Number analyzed (Eyes) | 9 | 5
Eyes | 7 | 5

ADVERSE EVENTS:
Time Frame: From baseline visit through 3 months of follow-up, the final study visit
Description: As mentioned previously in the results section, the number of eyes analyzed differs from the "started" row in Participant Flow Overview. Though 24 eyes were consented and met retention criteria, 6 eyes dropped out prior to complete baseline assessment and prior to surgery. Thus, there were 18 eyes "at risk" because only 18 eyes were operated on.
Arm/Group | DEXTENZA® Arm | Prednisolone Acetate 1% Arm
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 3/12 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DEXTENZA® Arm (N=12) | Prednisolone Acetate 1% Arm (N=6)
Eye pain with movement and lid twitching (Eye disorders) | 1 (1) | 0 (0) — Eye pain with movement and right upper lid twitching that occurred on post-op day 7 and resolved with supplemental topical anti-inflammatory eye drops.
Hyphema and shallow iris (Eye disorders) | 1 (1) | 0 (0) — 2mm hyphema and shallow iris that occurred on post-op day 1 and successfully resolved with topical atropine.
Floaters (Eye disorders) | 1 (1) | 0 (0) — New-onset small floaters that were noted by the patient on post-op day 30, likely unrelated to the surgery or intervention.

LIMITATIONS AND CAVEATS:
Early termination related to COVID-19 recruitment difficulties and loss to follow-up leading to small numbers of eyes analyzed. Length of follow-up limited to 3 months. Use of only three types of minimally invasive glaucoma surgery. Single-site, single-surgeon, open-label design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-18): https://cdn.clinicaltrials.gov/large-docs/51/NCT04200651/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT04200651/ICF_001.pdf